CLINICAL TRIAL: NCT00798135
Title: A Pilot Trial of Itraconazole Pharmacokinetics in Patients With Metastatic Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Kathy Miller, Ballvé-Lantero Professor of Medicine, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0809-10; IUCRO-0239
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Results first posted 2014-09-10 (Estimated); Last update posted 2023-12-21 (Actual); Status verified 2023-11

CONDITIONS: Breast Neoplasms; Neoplasm Metastasis
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- itraconazole (Experimental): Patients will receive oral itraconazole 200mg a day until disease progression.
  Interventions: Drug: itraconazole

INTERVENTIONS:
Drug: itraconazole — oral itraconazole 200mg a day until disease progression or unacceptable toxicities.

SUMMARY:
Cancer cells need to be able to make new blood vessels in order to keep growing. This is called angiogenesis. In a laboratory setting, the drug itraconazole was shown to help stop the growth of new blood vessels (anti-angiogenesis). It is hoped that itraconazole will prevent new blood vessels from forming in humans too.

The purpose of this study is to look at how the body processes and breaks down itraconazole (called pharmacokinetics). This study will also measure markers in your blood to see if itraconazole stops new blood vessels from forming. The safety of itraconazole will also be tested to see what effects (good and bad) it has on you and your breast cancer.

ELIGIBILITY:
Inclusion Criteria:

- Patients must have a pathologically confirmed diagnosis of invasive carcinoma of the breast. - Patients must carry a diagnosis of metastatic breast cancer. - Patients must be able to swallow oral medications. - Patients with HER 2+ tumors must have received trastuzumab in the past and may have had lapatinib. - Patients must have an ECOG performance status of 0-1. - Patients must be informed of the investigational nature of the study and must sign and give written informed consent. - Patients must have recovered to grade <1 from all acute toxicity of previous therapy for breast cancer with the exception of alopecia. - Adequate hematologic and hepatic function: 1)Absolute neutrophil count >= 1,500 mm3 2) Platelet count >= 100,000 mm3 3) Bilirubin <= 1.5mg/dL x ULN 4) AST and/or ALT <= 2 x ULN (< 5 x ULN in presence of known liver metastasis). - Prior to study enrollment, women of childbearing potential (WOCBP) must be advised of the importance of avoiding pregnancy during trial participation and must practice an effective method of birth control. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should also practice an effective method of birth control. - All WOCBP MUST have a negative serum or urine pregnancy test within 4 weeks prior to the start of study drug administration.

Exclusion Criteria:

* Use of the following concomitant medications within 14 days of starting protocol therapy is prohibited: Cisapride, dofetilide, ergot derivatives, levomethadyl, lovastatin, midazolam, pimozide, quinidine, simvastatin, or triazolam.
* Patients who are taking alprazolam (Xanax) are excluded from the trial.
* Patients must not have an active infection requiring the use of intravenous antibiotics. The use of oral antibiotics is allowed.
* Hypersensitivity to itraconazole, any component of the formulation, or to other azoles.
* Patients with uncontrolled CNS metastasis are excluded. If patients have CNS metastasis they must have completed brain radiation at least 2 weeks prior to registration and must be off steroids for CNS metastasis.
* Known preexisting congestive heart failure or left ventricular dysfunction. Patients with risk factors (ex. uncontrolled hypertension with BP >160/90) for cardiac dysfunction but no preexisting diagnosis of congestive heart failure or left ventricular dysfunction will have a screening EKG prior to enrollment. Subsequently, those patients with an abnormal EKG, as judged by the treating physician, will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-11; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Miller, MD, Principal Investigator — Indiana University Melvin and Bren Simon Cancer Center
Locations (1):
- Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Itraconazole
Started | 13
Completed | 0
Not Completed | 13
Not completed — Disease progression, relapse | 11
Not completed — Disease progression, refractory | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Itraconazole
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.8 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK) of Oral Itraconazole
Description: To determine the pharmacokinetics (PK) of oral itraconazole in patients with MBC by measuring mean trough plasma levels at steady state at weeks 2 and 4.
Time Frame: pre-dose at Weeks 2 and 4
Population: All patients with results available.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Itraconazole
Number analyzed (Participants) | 12
ng/mL
  Week 2 Intraconazole Concentration | 230.7 (216.8)
  Week 4 Intraconazole Concentration | 305.8 (334.8)
  Week 2 6-OH Itraconazole Concentration | 454.8 (429.3)
  Week 4 6-OH Itraconazole Concentration | 501.6 (502.6)

2. Secondary Outcome: Number of Patients With Adverse Events Grade 3 or 4 That Are Related to Study Treatment
Description: Number of patients with Adverse Events grade 3 or 4 that are related to study treatment. This will look into the safety of the study drug.
Time Frame: up to 100 months
Population: All patients in the study.
Measure: Number; unit: Participants
Arm/Group | Itraconazole
Number analyzed (Participants) | 13
Participants | 2

3. Secondary Outcome: Time to Progression.
Description: This is calculated as time till progression from treatment start until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months. If a patient did not progress, they were censored at the last evaluation visit. The median time till progression is calculated with its 95% confidence interval.
Time Frame: up to 100 months
Population: All patients in the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Itraconazole
Number analyzed (Participants) | 13
Months | 1.54 [0.89 to 2.73]

ADVERSE EVENTS:
Arm/Group | Itraconazole
Serious Adverse Events (participants affected / at risk) | 3/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Itraconazole (N=13)
NAUSEA (Gastrointestinal disorders) | 1 (1)
PAIN - ABDOMEN NOS (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
PAIN - BACK (Musculoskeletal and connective tissue disorders) | 1 (1)
HEMORRHAGE, GI - UPPER GI NOS (Gastrointestinal disorders) | 1 (1)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) - EXTREMITY-LOWER (Musculoskeletal and connective tissue disorders) | 1 (1)
PLEURAL EFFUSION (NON-MALIGNANT) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Itraconazole (N=13)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - SKIN (CELLULITIS) (Skin and subcutaneous tissue disorders) | 1 (1)
OCULAR/VISUAL (Eye disorders) | 1 (1)
VISION-BLURRED VISION (Eye disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 5 (5)
DIARRHEA (Gastrointestinal disorders) | 1 (1)
DISTENSION/BLOATING, ABDOMINAL (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL (Gastrointestinal disorders) | 1 (1)
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 1 (1)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) - ORAL CAVITY (Gastrointestinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 5 (5)
PAIN - ABDOMEN NOS (Gastrointestinal disorders) | 2 (2)
TASTE ALTERATION (DYSGEUSIA) (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 6 (6)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 3 (3)
PAIN (General disorders) | 1 (1)
BILIRUBIN (HYPERBILIRUBINEMIA) (Hepatobiliary disorders) | 1 (1)
ALKALINE PHOSPHATASE (Investigations) | 1 (1)
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 1 (1)
HEMOGLOBIN (Investigations) | 2 (2)
PLATELETS (Investigations) | 1 (1)
EDEMA: LIMB (Blood and lymphatic system disorders) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 4 (4)
PAIN - BACK (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN - BONE (Musculoskeletal and connective tissue disorders) | 2 (2)
PAIN - EXTREMITY-LIMB (Musculoskeletal and connective tissue disorders) | 2 (2)
PAIN - JOINT (Musculoskeletal and connective tissue disorders) | 1 (1)
INCONTINENCE, URINARY (Nervous system disorders) | 1 (1)
INSOMNIA (Nervous system disorders) | 1 (1)
INSOMNIA (Psychiatric disorders) | 4 (4)
NEUROPATHY: CRANIAL - CN VIII HEARING AND BALANCE (Nervous system disorders) | 1 (1)
NEUROPATHY: SENSORY (Nervous system disorders) | 2 (2)
PAIN - HEAD/HEADACHE (Nervous system disorders) | 1 (1)
SPEECH IMPAIRMENT (E.G., DYSPHASIA OR APHASIA) (Nervous system disorders) | 1 (1)
MOOD ALTERATION - ANXIETY (Psychiatric disorders) | 1 (1)
MOOD ALTERATION - DEPRESSION (Psychiatric disorders) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - PARANASAL (Respiratory, thoracic and mediastinal disorders) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - SINUS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
INFECTION WITH UNKNOWN ANC - SINUS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PAIN - CHEST WALL (Respiratory, thoracic and mediastinal disorders) | 1 (1)
URINARY FREQUENCY/URGENCY (Renal and urinary disorders) | 1 (1)
URINE COLOR CHANGE (Renal and urinary disorders) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS - URINARY TRACT NOS (Renal and urinary disorders) | 1 (1)
PAIN - BREAST (Reproductive system and breast disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 4 (4)
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY - NOSE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
VOICE CHANGES/DYSARTHRIA (E.G., HOARSENESS, LOSS OR ALTERATION IN VOICE, LARYNGITIS) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DERMATOLOGY/SKIN (Skin and subcutaneous tissue disorders) | 1 (1)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1)
HAIR LOSS/ALOPECIA (SCALP OR BODY) (Skin and subcutaneous tissue disorders) | 1 (1)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 1 (1)
RASH: ACNE/ACNEIFORM (Skin and subcutaneous tissue disorders) | 2 (2)
SWEATING (DIAPHORESIS) (Skin and subcutaneous tissue disorders) | 1 (1)
HOT FLASHES/FLUSHES (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes